CLINICAL TRIAL: NCT03934411
Title: Effect of Increased Pain Tolerance on Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Anti Doping Danmark (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Nikolai Nordsborg, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-17028397
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Opioid Use; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol treatment (Experimental)
  Interventions: Drug: Tramadol
- Placebo treatment (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tramadol — The subjects will orally ingest 100 mg tramadol retard actavis
  Arms: Tramadol treatment
Other: Placebo — The subjects will orally ingest 100 mg calcium powder
  Arms: Placebo treatment

SUMMARY:
Clinical prescription and use of opioids is a clear problem in large parts of the world and has the recent years received an increasing publicity in sports. This is in particular due to the World Anti-Doping Agency monitoring list, which reveal that endurance athletes utilize the opioid Tramadol frequently with the aim to enhance performance according to anecdotal evidence.

Studies investigating the effect of tramadol on exercise performance in healthy humans is limited to one study in moderate trained subjects. However, this effect may be different in highly trained subjects due to the effects of chronic exercise. Furthermore, ingestion of tramadol may impact motor-cognitive performance and it remains unknown whether tramadol can be detected in highly trained subjects following exercise.

In the present study the investigators apply a randomized double-blind placebo-controlled counterbalanced cross-over design to investigate whether tramadol treatment improves a preloaded cycling time trial performance, whether it affects motor-cognitive performance and whether it is detectable following exercise.

ELIGIBILITY:
Inclusion Criteria:

* Maximal oxygen uptake < 55 ml O2/min/kg
* Plasma creatinine concentration between 60-105 umol/L
* Plasma alanine aminotransferase between 10-70 U/L
* Familiarized with endurance training for at least a few years

Exclusion Criteria:

* Donated blood within the last 3 months
* Exposed to an altitude greater than 1000 m above sea level within the last two months
* Smoking

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Power output | 30 minutes
  Mean power output during a 15-km time trial
Motor-cognitive performance | 1 hour
  The motor-cognitive performance evaluated by mathematical calculations combined with the ability to pinch a certain force with the thumb and index finger
Detection rate | 1 day
  The detection rate of tramadol following the exercise intervention measured before, immediately after as well as 6 and 24h after treatment

SECONDARY OUTCOMES:
pH | 90 min
  The response of blood pH to exercise performance
Lactate | 90 min
  The response of blood lactate to exercise performance
Bicarbonate | 90 min
  The response of blood bicarbonate to exercise performance
Glucose | 90 min
  The response of blood glucose to exercise performance
Potassium | 90 min
  The response of blood potassium to exercise performance
Sodium | 90 min
  The response of blood sodium to exercise performance
Oxygen uptake | 90 min
  The response of systemic oxygen uptake during exercise performance
Pulmonary ventilation | 90 min
  The response of pulmonary ventilation during exercise performance.
Respiratory exchange ratio | 90 min
  The response of respiratory exchange ratio during exercise performance, calculated as the ratio between system oxygen uptake and systemic carbon monoxide production. The unit of measure is arbitrary.
Rate of Perceived Exertion | 90 min
  Measurement of the rate of perceived exertion by questionnaire during exercise performance using "The borg scale of perceived exertion", which range from 6 (minimum value) to 20 (maximum value). Higher values represent a higher perceived exertion.
Leg Pain | 90 min
  Measurement of the leg pain by questionnaire during exercise performance using the "10-point pain scale", which range from 0 (minimum) to 10 (maximum). Higher values represent a higher pain.
Heart rate | 90 min
  The response of heart rate to exercise performance
Power output during preload | 60 min
  Mean power output during a 60-min cycling exercise
Power output during time trial | 30 min
  The power output measured for each km of the time trial

OTHER OUTCOMES:
Height | 1 min
  Height of the subjects in cm
Weight | 1 min
  Weight of the subjects in kg
Age | 1 min
  Age of the subjects in years
Endurance training history | 1 min
  Endurance training history of subjects in years
Plasma creatinine | 10 min
  Concentration of plasma creatinine
Plasma alanine aminotransferase | 10 min
  Concentration of plasma alanine aminotransferase
Peak power of incremental test | 30 min
  The peak power of an incremental cycling test

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai B Nordsborg, Dr, Principal Investigator — Department of Nutrition, Exercise and Sports
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Denmark